CLINICAL TRIAL: NCT05065294
Title: An Open-Label Pilot Study Examining the Feasibility, Safety, and Effectiveness of Psilocybin Therapy for Depression in Bipolar II Disorder
Brief Title: Psilocybin Therapy for Depression in Bipolar II Disorder
Acronym: BAP
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Joshua Woolley, MD, PhD, Assistant Professor, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-32789
Record Dates: First submitted 2021-09-14; First posted 2021-10-04 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Bipolar II Disorder
Keywords: Bipolar; Depression; Psilocybin; Psychedelic; Psilocybin Therapy; Bipolar II; Safety
MeSH Terms: conditions — Bipolar Disorder; Depression

STUDY DESIGN:
Intervention Model Description: Open-label, single-arm, pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Psilocybin therapy (Experimental): Participants will receive one or two doses of psilocybin in a monitored setting approximately three weeks apart, with preparation sessions before and integration sessions after.
  Interventions: Drug: Psilocybin therapy

INTERVENTIONS:
Drug: Psilocybin therapy — - Psilocybin administration session 10mg-25mg delivered orally with psychological support and monitoring
  Other Names: 4-phosphoryloxy-N,N-dimethyltryptamine

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and feasibility of psilocybin therapy in people with Bipolar II Disorder.

DETAILED DESCRIPTION:
The primary goal of this study is to examine the safety, tolerability, and feasibility of psilocybin therapy in people with Bipolar II Disorder (BD II). Fourteen participants, ages 18 to 70 with clinically diagnosed BD II with active depression, in active outpatient mental health treatment, and who meet all other inclusion and exclusion criteria at screening will be enrolled. After baseline assessments, participants will engage in preparatory visits with trained facilitators, followed by an initial drug administration of oral psilocybin,supervised by the facilitators and a clinician who will conduct safety monitoring throughout. Participants will complete assessment and integration sessions with the facilitators subsequently in order to help process the experience. Participants who tolerated the first dosage may be asked to complete a second psilocybin dosing session, involving the same preparation, procedures, integration, and supervision as the first. Primary outcome measures will assess safety, tolerability, and feasibility of study procedures. Efficacy will be measured by change in depression as measured by the MADRS three weeks after the final psilocybin administration. Exploratory outcome measures will assess changes in sleep, quality of life, and therapeutic engagement.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70
* Comfortable speaking and writing in English
* Diagnosis of Bipolar Disorder II with current depression
* Have a care partner/support person available throughout the study
* Able to attend all in-person visits at UCSF as well as virtual visits
* Having tried at least one previous medication trials for their bipolar disorder, each lasting at 6 weeks or more.

Exclusion Criteria:

* Current or previous diagnosis of Bipolar I Disorder
* History of schizophrenia spectrum or psychotic disorder
* Use of psychedelics within the past 6 months, including MDMA
* Current diagnosis of cancer
* Seizures that continue to the present
* Fear of blood or needles
* Regular use of medications that may have problematic interactions with psilocybin, including but not limited to antidepressants (Bupropion allowed), serotonin antagonists, some antipsychotics, dopamine agonists/antagonists, stimulants, opioids, and Lithium.
* A health condition that makes this study unsafe or unfeasible, determined by study physicians

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2022-01-28 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of psilocybin therapy for depression in BD II | Baseline to 3 months following last drug dose
  -Incidence, severity, and frequency of Adverse Events (AEs) including Treatment-Emergent AEs (TEAEs) and Serious AEs (SAEs)
Recruitment rate | Baseline to 3 months following last drug dose
  -Measured as a percentage of participants who were contacted for pre-screening and consented.
Retention rate | Baseline to 3 months following last drug dose
  -Measured as a percentage of participants who began and completed treatment.
Clinician-reported effects of psilocybin therapy on depressive symptoms in people with Bipolar II | Baseline to 3 weeks following last drug dose
  * Montgomery-Asberg Depression Rating Scale (MADRS)
  * Each item is scored on a on a scale of 0-6 with a total score of 0-60
  * Higher scores correspond to worse outcomes
Treatment Satisfaction of study procedures | Baseline to 3 months following last drug dose
  * Measured by the treatment satisfaction questionnaire
  * 5-item scale, plus three free response questions
  * Higher scores representing better treatment satisfaction
Self-reported effects of psilocybin therapy on manic and/or psychotic symptoms in people with Bipolar II | Baseline to 11 days following each drug dose
  * Altman Self-Rating Mania Scale(ASRM-14)
  * Each item rated on a 0 to 4 scale, with a total score of 0 to 56
  * Higher scores indicating greater severity of manic symptoms, with items that also measure psychosis
Clinician-reported effects of psilocybin therapy on mania symptoms in people with Bipolar II | Baseline to 3 months following each drug dose
  * Young Mania Scale(YMS)
  * 7 items are rated on a 0 to 4 scale and 4 items are rated on a 0 to 8 scale. The total score ranges from 0-60
  * Higher scores indicating greater severity of manic symptoms.
Clinician-reported effects of psilocybin therapy on suicidality symptoms in people with Bipolar II | Baseline to 3 months following last drug dose
  * Columbia-Suicide Severity Rating Scale (C-SSRS)
  * Characterizes suicidal ideation in three separate categories with a total score range from 0-25
  * Higher scores indicate greater severity

SECONDARY OUTCOMES:
Patient reported effects of psilocybin therapy on depressive symptoms symptoms in people with Bipolar II (exploratory) | Baseline to 3 months following last drug dose
  * Quick Inventory of Depressive Symptomatology (QIDS-SR)
  * Each item is scored on a on a scale of 0-3, with a total score of 0-27
  * Higher scores correspond to worse outcomes
Effects of psilocybin therapy on anxiety symptoms in people with Bipolar II (exploratory) | Baseline to 3 months following last drug dose
  * Generalized Anxiety Disorder 7-item scale (GAD-7)
  * Each item is rated on a scale from 0-3, with a total score of 0-21
  * Higher scores correspond to worse outcomes
Effects of psilocybin therapy on sleep quality in people with Bipolar II (exploratory) | Baseline to 3 months following last drug dose
  * Insomnia Severity Index (ISI)
  * Each item is scored on a scale of 0-4 with a total score range of 0-28
  * Higher scores indicate greater severity in sleep disturbance
Effects of psilocybin therapy on quality of life in people with Bipolar II (exploratory) | Baseline to 3 months following last drug dose
  * Quality of Life in Bipolar Disorder Questionnaire (QoL-BD)
  * Each item is scored on a scale of 1-5 with a total score range of 48-240
  * Higher scores indicate greater quality of life
Effects of psilocybin therapy on borderline personality disorder symptoms in people with Bipolar II (exploratory) | Baseline to 3 months following last drug dose
  * Zanarini Rating Scale (ZRS)
  * Each item is scored on a scale of 0-4 with a total score range of 0-30
  * Higher scores indicate greater severity in symptoms
Effects of psilocybin therapy on adult attachment in people with Bipolar II (exploratory) | Baseline to 3 months following last drug dose
  * Experiences in Close Relationships-Modified 16-Item Scale (ECR-M16)
  * Each item is scored on a scale of 1-7 with a total score range of 8-126
  * Lower scores on each dimension of attachment anxiety and avoidance represent greater levels of attachment security
Effects of psilocybin therapy on participant-reported recovery in people with Bipolar II (exploratory) | Baseline to 3 months following last drug dose
  * Bipolar Recovery Questionnaire (BRQ)
  * 36 items (visual analog scales)
  * Higher total scores indicate a higher degree
Subjective effects of psilocybin therapy in people with Bipolar II | Baseline to 3 months following last drug dose
  * 5-Dimensional Altered States of Consciousness Rating Scale (5D-ASC)
  * 94 items (visual analog scales) broken down into subcategories to quantify the acute subjective effects of psilocybin directly following each psilocybin administration session
Subjective effects of psilocybin therapy in people with Bipolar II | 3 weeks following last drug dose
  * Study specific Transformational Experiences Questionnaire (TEQ)
  * Meant to quantify subjective effects of psilocybin on 1-7 scale

CONTACTS AND LOCATIONS:
Overall Officials: Joshua D Woolley, MD,PhD, Principal Investigator — University of California, San Francisco; David Guard, PhD, Study Director — San Francisco State University
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grande I, Berk M, Birmaher B, Vieta E. Bipolar disorder. Lancet. 2016 Apr 9;387(10027):1561-1572. doi: 10.1016/S0140-6736(15)00241-X. Epub 2015 Sep 18. PMID 26388529
- [Background] Carhart-Harris RL, Bolstridge M, Rucker J, Day CM, Erritzoe D, Kaelen M, Bloomfield M, Rickard JA, Forbes B, Feilding A, Taylor D, Pilling S, Curran VH, Nutt DJ. Psilocybin with psychological support for treatment-resistant depression: an open-label feasibility study. Lancet Psychiatry. 2016 Jul;3(7):619-27. doi: 10.1016/S2215-0366(16)30065-7. Epub 2016 May 17. PMID 27210031
- [Background] Carhart-Harris RL, Bolstridge M, Day CMJ, Rucker J, Watts R, Erritzoe DE, Kaelen M, Giribaldi B, Bloomfield M, Pilling S, Rickard JA, Forbes B, Feilding A, Taylor D, Curran HV, Nutt DJ. Psilocybin with psychological support for treatment-resistant depression: six-month follow-up. Psychopharmacology (Berl). 2018 Feb;235(2):399-408. doi: 10.1007/s00213-017-4771-x. Epub 2017 Nov 8. PMID 29119217
- [Background] Griffiths RR, Johnson MW, Carducci MA, Umbricht A, Richards WA, Richards BD, Cosimano MP, Klinedinst MA. Psilocybin produces substantial and sustained decreases in depression and anxiety in patients with life-threatening cancer: A randomized double-blind trial. J Psychopharmacol. 2016 Dec;30(12):1181-1197. doi: 10.1177/0269881116675513. PMID 27909165
- [Background] Szmulewicz AG, Angriman F, Samame C, Ferraris A, Vigo D, Strejilevich SA. Dopaminergic agents in the treatment of bipolar depression: a systematic review and meta-analysis. Acta Psychiatr Scand. 2017 Jun;135(6):527-538. doi: 10.1111/acps.12712. Epub 2017 Mar 3. PMID 28256707